CLINICAL TRIAL: NCT01288677
Title: Phase I, First In-human, Double-blind, Randomized, Placebo-controlled Trial to Examine the Safety, Tolerability, and Blood and Plasma Pharmacokinetics of Increasing Single Oral Doses of TMC649128
Brief Title: TMC649128HPC1001 - First In-human Trial to Examine Safety, Tolerability, and Pharmacokinetics (How the Drug is Absorbed Into the Bloodstream) of Increasing Single Oral Doses of TMC649128 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: CR017272; TMC649128HPC1001 (Other: Tibotec Pharmaceuticals)
Record Dates: First submitted 2011-01-13; First posted 2011-02-02 (Estimated); Last update posted 2013-03-20 (Estimated); Status verified 2013-03

CONDITIONS: Healthy Volunteer
Keywords: Healthy volunteer; TMC649128HPC1001; TMC649128; HCV; Hepatitis C; healthy volunteers; Phase I trial
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (1):
- 001 (Experimental): TMC649128 Escalated doses
  Interventions: Drug: TMC649128

INTERVENTIONS:
Drug: TMC649128 — Escalated doses

SUMMARY:
The purpose of this study is to assess the pharmacokinetics, safety, and tolerability of single oral doses of TMC649128 in healthy volunteers. Pharmacokinetics (PK) means how the drug is absorbed into the bloodstream, distributed in the body, and eliminated from the body.

DETAILED DESCRIPTION:
TMC649128 will be investigated for the treatment of chronic hepatitis C infection. This is a Phase I, first in humans (no clinical studies have been performed to date), double-blind (neither the participant nor investigator knows whether they receive active or placebo), randomized (study medication is assigned by chance), placebo-controlled study to examine the safety, tolerability, and blood and plasma pharmacokinetics of increasing single oral doses of TMC649128. The single dose escalation will consist of 6 sessions (Sessions I to IV) in 6 panels (Panels 1 to 6) of 9 healthy adult volunteers each. The dose of TMC649128 will be consecutively escalated. In each session, 6 participants will receive TMC649128 and 3 participants will receive placebo, all with standard meals. Each session will have a staggered approach, ie, the first 4 participants will be dosed, followed by at least a 72-hour safety review and if no acute effects are observed, the remaining 5 participants will be dosed. The main focus of the trial is the determination of safety and tolerability of TMC649128 after single oral doses in fed conditions in healthy volunteers, but also the determination of the pharmacokinetic characteristics (level-profile of TMC649128 over time in the blood stream and urine). This evaluation requires multiple blood samples from Day 1 to Day 4. Safety assessments (blood and urine tests, blood pressure, pulse, electrocardiogram, and physical examination) will follow a different schedule and will be performed during each session, up to 4 weeks after the last administration. Safety and tolerability evaluations will be recorded at regular intervals throughout the trial. The single dose escalation will consist of 6 sessions in 6 panels of 9 healthy adult volunteers each. The dose of TMC649128 will be consecutively escalated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy based on a medical evaluation including medical history, physical examination, blood tests and electrocardiogram
* Body Mass Index of 18.0 to 30.0 kg/m² and non-smoker for at least 3 months prior to selection
* Women must be postmenopausal for at least 2 years and/or be surgically sterile.

Exclusion Criteria:

* Infection with Hepatitis A, B or C virus
* infection with the Human Immunodeficiency Virus (HIV)
* History of, or any current medical condition which could impact the safety of the participant in the study
* A positive urine drug test at screening
* History of any drug allergy or clinically relevant skin disease
* Participation in an investigational drug trial or received an investigational vaccine within 30 days prior to intake.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2011-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Number of volunteers with adverse events, if any | Up to Day 4
Laboratory evaluations of blood and urine samples | Up to Day 4
Vital signs evaluations | Up to Day 4
Electrocardiogram evaluations | Up to Day 4

SECONDARY OUTCOMES:
Plasma concentration of TMC649128 after a single oral dose of TMC649128 in healthy volunteers in fed conditions | Measured on Day 1 to Day 4

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Clinical Trial, Study Director — Tibotec Pharmaceutical Limited